CLINICAL TRIAL: NCT02823561
Title: Efficacy and Tolerability of Garcinia Mangostana Extracts in the Management of Weight Loss in Severe Obese Patients
Brief Title: Garcinia Mangostana Extracts in the Management of Weight Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Carla Lubrano, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URomLS-01
Record Dates: First submitted 2016-06-23; First posted 2016-07-06 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-06

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Garcinia mangostana (treatment group) (Active Comparator): Balanced low-calorie diet and regular exercise in combination with integration
  Interventions: Dietary Supplement: Garcinia mangostana
- Control group (Other): balanced low-calorie diet and regular exercise
  Interventions: Behavioral: Control group

INTERVENTIONS:
Dietary Supplement: Garcinia mangostana
  Arms: Garcinia mangostana (treatment group)
Behavioral: Control group
  Arms: Control group

SUMMARY:
Obesity is one of the greatest public health challenges of the 21st century. Its prevalence has tripled in many countries of the European Region since the 1980s, and the numbers of those affected continue to rise at an alarming rate. In addition to causing various physical disabilities and psychological problems, excess weight drastically increases a person's risk of developing a number of noncommunicable diseases including cardiovascular disease, cancer and diabetes, in association or not to metabolic syndrome. The risk of developing more than one of these diseases (co-morbidity) also increases with increasing body weight. Every year a growing number of patient tend to suffer of more severe obesity and difficulty in losing weight even with a restricted diet and exercise.

Garcinia mangostana (Sphaeranthus indicus extract) has known for its antioxidant properties; new evidence point out some promising effects in the prevention of lipogenesis and the promotion of lipolysis . Currently in the scientific literature there is only one paper, by Stern et al., showing the association of Garcinia mangostana assumption in low-calorie diet. This work has demonstrated a significant reduction in weight loss , compared to the placebo group,due to the use of Garcinia mangostana.

Aim of the present study is the evaluation of safety and efficacy of weight loss in severe obese patients. Also cardiometabolic parameters and flogosys serum indicators will be evaluated before and after 6 month therapy of low calory diet alone or in association with Garcinia mangostana extract.

DETAILED DESCRIPTION:
After the screening visit for the evaluation of the inclusion / exclusion criteria and sign informed consent(Visit 1), each patient will be randomized (Visit 2; Time 0; Baseline) (1: 1) to receive two different treatment for the duration of 26 weeks:

1. low-calorie balanced diet consistent exercise (control group)
2. balanced low-calorie diet and regular exercise in combination with the assumption of Garcinia mangostana (treatment group)

Throughout the duration of the study, every eight weeks, unless otherwise indicated from the specialists, for each subject was expected a nutritional and an endocrinological visit with a anthropometric parameter check (body composition) and compliance to therapy (dietary / physical activity diary).

Also a bood sample test was performed to evaluate electrocardiogram, lipid profile, glucose tolerance, hormonal parameters, inflammatory and bone markers.

ELIGIBILITY:
Inclusion Criteria:

* Obesity: BMI >35 kg/m2.
* Stable medical therapy for comorbidities from at least 6 months

Exclusion Criteria:

* Hormonal replacement therapy
* Hyperprolactinaemia and /or other endocrine hypothalamic-pituitary diseases (empty sella syndrome and expansive pituitary disorders evaluated by MRI)
* Any other condition that medical judgment precludes patient safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Weight loss - Kg reduction | 26 weeks

SECONDARY OUTCOMES:
Insulin sensitivity assessed by the homeostatic model assessment (HOMA-IR) | 26 weeks
Lipid profile by serum biochemistry | 26 weeks
Abdominal obesity measured by waist circumference | 26 weeks
Body composition by Dexa parameters | 26 weeks
Changes in microalbuminuria by unin analysis | 26 weeks

IPD SHARING:
Plan to Share IPD: No